CLINICAL TRIAL: NCT01134094
Title: Combined Randomised and Observational Study of Type B Ankle Fracture Treatment
Acronym: CROSSBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: CROSSBAT Investigators (Unknown)
Responsible Party: Principal Investigator, Rajat Mittal, Principal Investigator, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROSSBAT
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Ankle Fractures
Keywords: Undisplaced; Ankle Fracture; Weber B
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Operative (Active Comparator): Patients who are treated non-operatively will be treated with a walking boot and allowed WBAT. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. All patients will be reviewed between 7 and 14 days post injury with repeat x-rays by the treating surgeon.
  Interventions: Procedure: Non Operative
- Operative (Active Comparator): The specific procedure for each patient managed operatively, both in the observational study and the RCT, will be determined by the operating surgeon. Any adverse intra-operative or post-operative event will be recorded. This includes but is not limited to death, infection and neurovascular injury. Post operatively, all patients will be NWB (non weight bearing) and placed in a POP (plaster of paris) below knee cast or walking boot. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. The treating surgeon will review the patients after 10-14 days for a wound review, removal of sutures and change of cast to a fibreglass cast or walking boot (cam walker). The patient will be WBAT (weight bearing as tolerated) for a further 4 weeks.
  Interventions: Procedure: Open reduction internal fixation of the ankle

INTERVENTIONS:
Procedure: Open reduction internal fixation of the ankle — The specific procedure for each patient managed operatively, both in the observational study and the RCT, will be determined by the operating surgeon. Any adverse intra-operative or post-operative event will be recorded. This includes but is not limited to death, infection and neurovascular injury. Post operatively, all patients will be NWB (non weight bearing) and placed in a POP (plaster of paris) below knee cast or walking boot. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. The treating surgeon will review the patients after 10-14 days for a wound review, removal of sutures and change of cast to a fibreglass cast or walking boot (cam walker). The patient will be WBAT (weight bearing as tolerated) for a further 4 weeks.
  Arms: Operative
Procedure: Non Operative — Patients who are treated non-operatively will be treated with a walking boot and allowed WBAT. Discharge from hospital will be determined by the patient walking 25m unaided by standby assistance. All patients will be reviewed between 7 and 14 days post injury with repeat x-rays by the treating surgeon.
  Arms: Non-Operative

SUMMARY:
This study will determine whether operative management confers improved short and long-term outcomes for patients with isolated AO type 44-B1 distal fibula fractures when compared with non-operative management.

DETAILED DESCRIPTION:
Background:

Ankle fractures are common. Recent clinical studies have shown that there is an increasing incidence of ankle fractures. Treatments vary and there is no clear consensus of the ideal approach to type 44-B1 distal fibular fractures. They range from open reduction and internal fixation to restore anatomical alignment to wearing below-knee walking plaster for an average of six weeks.

The argument for surgical fixation is that it addresses minor displacement and possible future displacement therefore potentially preventing future arthritis. On the other hand, there are numerous complications associated with surgery.

The argument for non-operative treatment is that non-union is not a common complication. Therefore surgery can be avoided in the majority of cases avoiding the clinical risks associated with surgery.

Aim:

Primary aim: To compare, ankle function and quality of life in the 12 months following an isolated AO type 44-B1 distal fibula fracture minimal talar shift, between patients treated operatively and non-operatively.

Secondary aims:

1. To compare the recovery of ankle function and quality of life between the two study groups from 3 months to 1 year post ankle fracture
2. To compare complications between the two groups.
3. To conduct a health economic analysis between the two groups as indicated

Research Design: Combined Randomised and Observational Study

Methods:

Recruitment:

All consecutive patients who present to a recruiting hospital with a distal fibular fracture during the study period will be screened for eligibility. In most hospitals, all surgeons on the on-call roster will participate in the study. Consenting patients of the surgeons who have agreed to participate in the randomised arm of the trial will be invited to have their treatment randomised. Patients of surgeons involved in the observational component of the study will be invited to be included in the observational arm together with the patients who decline to be randomised, but consent to follow-up

Written, informed consent will be obtained.

Eligible patients of surgeons participating in the randomised arm will have the option of having their treatment randomised. If consent is given, the surgeon will call a central number for patient allocation that is available 24 hours per day, 7 days per week. The randomisation schedule will be prepared and administered by an external party not otherwise involved in the study. If the patient declines randomisation, treatment will be determined after surgeon-patient discussion. Eligible patients of surgeons involved in the observational arm will also have their treatment provided (operative or non-operative) as per usual surgeon practice.

Typical demographic, anthropometric and surgical details (where appropriate) will be recorded for contextual reference.

Surgical intervention:

The surgical technique for each patient managed operatively, in both the observational and randomised arms of the study, will include fixation using a plate and screws. Any adverse intra-operative or post-operative event will be recorded. This includes but is not limited to death, infection, VTE and neurovascular injury. Post-operatively, all patients will be non weight bearing and placed in a below-knee plaster cast or walking boot. Discharge from hospital will be determined by the patient's ability to walk 25 m unaided by standby assistance as determined by a physiotherapist. The treating surgeon will review the patient after 10-14 days for assessment of the wound, removal of sutures and change of cast to a fibreglass cast or walking boot (cam walker). The patient will then be allowed to WBAT (weight bearing as tolerated) for a further 4 weeks. This protocol represents usual post-operative practice for this injury, as determined through meetings with the Australian Orthopaedic Trauma Society.

Non-Operative management:

Patients who are treated non-operatively will be treated with a walking boot and allowed WBAT. Discharge from hospital will be determined as for the surgical arm. All patients will be reviewed between 7 and 14 days post injury with repeat radiographs by the treating surgeon. This represents usual non-operative treatment for this injury.

Other management decisions such as need for antibiotics, VTE prophylaxis or anaesthetic type will be as per usual care for that institution and recorded by the research team. Referral for further physiotherapy post removal of cast or boot (either study arm) will be based on the presence of overt ankle stiffness affecting gait. The use of physiotherapy (type and duration) will be noted. Specific prescription of the type of physiotherapy is not possible as patients will be free to access public and private services. Study participants will record all hospitalisations and visits to any health professional. They will be required to report the main reason for such health service occasions during the first year of follow-up period.

Outcomes will be collected and results will be reported in peer-reviewed journals after appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Arbeitsgemeinschaft für Osteosynthesefragen (AO) type 44-B1 fibula fracture
* Patients aged between 18 and 65 inclusive.
* No talar shift - Medial clear space less than 2mm compared with the superior clear space on anterior-posterior (AP) view of the ankle.
* Closed injury
* No concurrent fractures/dislocations
* Mobilising unaided/independently pre-injury
* Willingness to be followed up for 12 months
* Able to provide informed written consent

Exclusion Criteria:

* Medically fit for general anaesthesia/surgery
* Dislocation on presentation
* Skeletally immature patients
* Previous trauma or surgery to the affected ankle
* Pregnancy
* Other injuries that impede mobilisation e.g. stroke, neurovascular deficit at presentation
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
American Academy of Orthopaedic Surgeons Foot and Ankle Questionnaire | 12 months
  American Academy of Orthopaedic Surgeons Foot and Ankle Outcomes Questionnaire
PCS of Short Form (SF)-12v2 | 12 months
  SF-12 version 2 Health Survey

SECONDARY OUTCOMES:
Complications | 6 weeks, 3, 6 and 12 months
  Late surgery Infection Neurovascular complication Mortality
American Academy of Orthopaedic Surgeons (AAOS) Foot and Ankle Questionnaire | 3 and 6 months
  American Academy of Orthopaedic Surgeons (AAOS) Foot and Ankle Questionnaire
MCS of Short Form (SF)-12v2 | 3, 6 and 12 months
  Short Form (SF)-12v2
PCS Short Form (SF)-12v2 | 3 and 6 months
  Short Form (SF)-12v2

CONTACTS AND LOCATIONS:
Overall Officials: Ian Harris, MBBS, PhD, FRACS, Principal Investigator — University of New South Wales, Whitlam Orthopaedic Research Centre; Rajat Mittal, Bsc (Med) MBBS, Principal Investigator — University of New South Wales, Whitlam Orthopaedic Research Centre
Locations (21):
- Australia (21):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Brisbane and Women's Hospital, Brisbane, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Royal Prince Alfred, Camperdown, New South Wales
  - Sutherland Hospital, Caringbah, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - The Alfred Hospital, Melbourne, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - The Royal Melbourne Hospital, Parkville, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Cairns Base Hospital, Cairns, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - Nambour Hospital, Nambour, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Mittal R, Harris IA, Adie S, Naylor JM; CROSSBAT Study Group. Surgery for Type B Ankle Fracture Treatment: a Combined Randomised and Observational Study (CROSSBAT). BMJ Open. 2017 Mar 27;7(3):e013298. doi: 10.1136/bmjopen-2016-013298. PMID 28348185